CLINICAL TRIAL: NCT03464526
Title: A Double-Blind, Randomised, Placebo Controlled Study of the Efficacy and Safety and Pharmacokinetics of Orvepitant in Subjects With Pruritus Associated With Atopic Dermatitis
Brief Title: A Study of the Efficacy and Safety of Orvepitant in Subjects With Pruritus Associated With Atopic Dermatitis
Acronym: SOOTHE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORV-ADP-01
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Pruritus; Atopic Dermatitis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic | interventions — orvepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orvepitant 10mg (Active Comparator): Orvepitant 10mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant
- Orvepitant 20mg (Active Comparator): Orvepitant 20mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant
- Orvepitant 30mg (Active Comparator): Orvepitant 30mg tablet, once daily for 12 weeks
  Interventions: Drug: Orvepitant
- Placebo (Placebo Comparator): Placebo tablet, once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orvepitant — Tablet, once daily, oral
  Arms: Orvepitant 10mg; Orvepitant 20mg; Orvepitant 30mg
Drug: Placebo — Tablet, once daily, oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of three doses of orvepitant, taken once a day, in the treatment of pruritus associated with atopic dermatitis.

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, parallel group, placebo-controlled dose range study in subjects with pruritus associated with atopic dermatitis.

Doses of orvepitant (10 mg/day, 20 mg/day and 30 mg/day) and placebo will be investigated in four parallel groups.

Each group will compromise of approximately 100 subjects, randomized 1:1:1:1 (approximately 400 subjects in total).

All subjects will enter a two-week screening period to determine eligibility. Eligible subjects will be randomized at the Baseline/Day 1 visit and enter a 12-week double-blind dosing period. During this period there will be four visits at Weeks 2, 4, 8 and 12. There will be a final safety follow-up visit four weeks after the end of the treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of Atopic Dermatitis for ≥ 6 months confirmed by either the UK Working Party definition or the Hanifin definition
* Subjects must have chronic (> 6 months) pruritus which is unresponsive or inadequately responsive to current therapies such as topical steroids or antihistamines
* Subjects must have atopic dermatitis with a severity > 3 on the IGA and EASI ≥12 at Screening visit/Visit 1

Key Exclusion Criteria:

* Presence of, or history of, any other inflammatory dermatosis or skin conditions which may cause pruritus
* Any other possible cause for pruritus eg systemic, neurological, idiopathic, or metabolic
* Acute super-infection of AD lesions requiring treatment with antibiotics within 4 weeks of Visit 2
* Inability to comply with the use of prohibited and allowed medications as described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in Itch Intensity - Numeric Rating Scale | Week 12
  Change from baseline in the mean worst NRS pruritus intensity scores recorded by the subject during the last 3 days of available values in the period prior to the week 12 visit

IPD SHARING:
Plan to Share IPD: No